CLINICAL TRIAL: NCT04948333
Title: A Phase 3b, Multi-center, Open-label, Treatment Optimization Study of Oral Asciminib in Patients With Chronic Myelogenous Leukemia in Chronic Phase (CML-CP) Previously Treated With 2 or More Tyrosine Kinase Inhibitors
Brief Title: Asciminib Treatment Optimization in ≥ 3rd Line CML-CP
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CABL001A2302; 2024-511381-36-00 (EU CTIS Number: EU CT number)
Record Dates: First submitted 2021-06-28; First posted 2021-07-01 (Actual); Results first posted 2025-03-27 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Chronic Myelogenous Leukemia
Keywords: ABL001; Phase 3; tyrosine kinase inhibitor; Chronic myelogenous leukemia (CML); chronic myeloid leukemia (CML); chronic myelocytic leukemia (CML); chronic granulocytic leukemia (CGL); cancer of the white blood cells; clonal bone marrow stem cell disorder; proliferation of mature granulocytes; Treatment optimization; Asciminib; European Leukemia Network (ELN) Recommendations 2020; Major Molecular Response (MMR) rate at 48 weeks
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — asciminib; BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ABL001 (Experimental): Participants will be treated with 80 mg of ABL001 (40 mg BID or 80mg QD). In patients not achieving MMR at 48 weeks or losing the response after the week 48 assessment up to week 108, asciminib dose may be escalated to 200 mg q.d. if in the investigator's opinion the patient may benefit from the escalation.
  Interventions: Drug: ABL001 40mg BID; Drug: ABL001 80mg QD; Drug: ABL001 200mg QD

INTERVENTIONS:
Drug: ABL001 40mg BID — One tablet of 40 mg will be taken orally twice a day (BID)
  Other Names: asciminib
Drug: ABL001 80mg QD — Two tablets of 40 mg will be taken orally once a day (QD)
  Other Names: asciminib
Drug: ABL001 200mg QD — Five tablets of 40 mg will be taken orally once a day (QD)
  Other Names: asciminib

SUMMARY:
The purpose of the study is to optimize the treatment of asciminib in patients with chronic myelogenous leukemia in chronic phase (CML-CP) previously treated with 2 or more Tyrosine Kinase Inhibitors (TKIs).

DETAILED DESCRIPTION:
This study consists of a screening period of up to 28 days, a treatment period of 144 weeks and a post-treatment safety follow-up period of 4 weeks.

Patients will receive asciminib as study treatment continuously for up to 144 weeks or until disease progression, treatment failure or intolerance to treatment. At treatment initiation, asciminib will be provided to all trial patients at a total daily dose of 80 mg. All patients will be randomly assigned 1:1 to 2 groups with 80 mg given either as 40 mg b.i.d. or 80 mg q.d., using IRT to avoid any selection bias.

In patients not achieving Major Molecular Responses (MMR) at 48 weeks or losing the response after the week 48 assessment up to week 108, asciminib dose may be escalated to 200 mg q.d. if in the investigator's opinion the patient may benefit from the escalation. In addition, there must not be any grade 3 or 4 toxicity while on therapy, or persistent grade 2 toxicity, possibly related to asciminib and unresponsive to optimal management.

The trial will enroll a total of approximately 186 patients:

* 156 patients with CML-CP not in MMR at baseline who were treated with two or more TKIs and who were either resistant (ELN 2020 warning or failure) or intolerant to the last treatment will be enrolled. For this population, the primary endpoint for MMR at 48 weeks will be assessed.
* Up to 30 additional patients intolerant only to their last TKI treatment and in MMR at baseline will also be enrolled. This patient population will not be part of primary endpoint analysis; however, all assessments will be done as with the 156 patients from the population of the primary endpoint analysis.

ELIGIBILITY:
Key Inclusion criteria:

* Signed informed consent must be obtained prior to participation in the study
* Male or female patients with a diagnosis of CML-CP ≥ 18 years of age
* Treatment with a minimum of 2 or more prior TKIs (i.e. imatinib, nilotinib, dasatinib, bosutinib, radotinib or ponatinib)
* Warning or failure (adapted from the 2020 ELN Recommendations) or intolerance to the most recent TKI therapy at the time of screening
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1, or 2
* Adequate end organ function (as per central laboratory tests)

Key Exclusion criteria:

* Known presence of the BCR::ABL1 T315I mutation at any time prior to study entry
* Known second chronic phase of CML after previous progression to AP/BC
* Previous treatment with a hematopoietic stem-cell transplantation
* Patient planning to undergo allogeneic hematopoietic stem cell transplantation
* Uncontrolled cardiac repolarization abnormality
* Severe and/or uncontrolled concurrent medical disease that in the opinion of the investigator could cause unacceptable safety risks or compromise compliance with the protocol
* History of acute pancreatitis within 1 year of study entry or past medical history of chronic pancreatitis
* Testing for Hepatitis B surface antigen (HbsAg) and Hepatitis B core antibody (HBcAb / anti HBc) will be performed at screening. Patients with active Hepatitis B Virus (HBV) infection (hepatitis B surface antigen [HbsAg] positive) will be excluded

Other Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2026-02-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (46):
- Argentina (2):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Buenos Aires
- Austria (3):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Vienna
- Brazil (2):
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, São Paulo
- Canada (2):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Toronto, Ontario
- France (5):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
- Germany (6):
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Jena, Thuringia
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, München
- Greece (2):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Thessaloniki
- Italy (3):
  - Novartis Investigative Site, Monza, MB
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Verona, VR
- Malaysia (4):
  - Novartis Investigative Site, George Town, Pulau Pinang
  - Novartis Investigative Site, Kota Kinabalu, Sabah
  - Novartis Investigative Site, Johor Bahru
  - Novartis Investigative Site, Kuala Selangor
- Novartis Investigative Site, Khoudh, Oman
- Poland (2):
  - Novartis Investigative Site, Katowice
  - Novartis Investigative Site, Warsaw
- Novartis Investigative Site, Singapore, Singapore
- South Korea (3):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
  - Novartis Investigative Site, Taegu
- Spain (5):
  - Novartis Investigative Site, Santiago Compostela, A Coruna
  - Novartis Investigative Site, Bilbao, Bizkaia
  - Novartis Investigative Site, Santa Cruz, Santa Cruz De Tenerife
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
- United Kingdom (3):
  - Novartis Investigative Site, Leeds, West Yorkshire
  - Novartis Investigative Site, Cambridge
  - Novartis Investigative Site, London
- Vietnam (2):
  - Novartis Investigative Site, Hanoi
  - Novartis Investigative Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study is conducted globally across 16 countries.
Groups:
- Asciminib 40 mg b.i.d. - Subjects Without MMR at Baseline: Asciminib 40 mg b.i.d. - Subjects without MMR at baseline: Participants will be treated with 80 mg of ABL001 (40 mg BID). In patients not achieving MMR at 48 weeks or losing the response after the week 48 assessment up to week 108, asciminib dose may be escalated to 200 mg q.d. if in the investigator's opinion the patient may benefit from the escalation.
- Asciminib 80 mg q.d. - Subjects Without MMR at Baseline: Asciminib 80 mg q.d. - Subjects without MMR at baseline: Participants will be treated with 80 mg of ABL001 (80mg QD). In patients not achieving MMR at 48 weeks or losing the response after the week 48 assessment up to week 108, asciminib dose may be escalated to 200 mg q.d. if in the investigator's opinion the patient may benefit from the escalation.
- Asciminib 40 mg b.i.d. - Subjects With MMR at Baseline: Asciminib 40 mg b.i.d. - Subjects with MMR at baseline: Participants will be treated with 80 mg of ABL001 (40 mg BID). In patients not achieving MMR at 48 weeks or losing the response after the week 48 assessment up to week 108, asciminib dose may be escalated to 200 mg q.d. if in the investigator's opinion the patient may benefit from the escalation.
- Asciminib 80 mg q.d. - Subjects With MMR at Baseline: Asciminib 80 mg q.d. - Subjects with MMR at baseline: Participants will be treated with 80 mg of ABL001 (80mg QD). In patients not achieving MMR at 48 weeks or losing the response after the week 48 assessment up to week 108, asciminib dose may be escalated to 200 mg q.d. if in the investigator's opinion the patient may benefit from the escalation.
Period: Overall Study
Arm/Group | Asciminib 40 mg b.i.d. - Subjects Without MMR at Baseline | Asciminib 80 mg q.d. - Subjects Without MMR at Baseline | Asciminib 40 mg b.i.d. - Subjects With MMR at Baseline | Asciminib 80 mg q.d. - Subjects With MMR at Baseline
Started | 85 | 84 | 14 | 16
Full Analysis Set (FAS) (All subjects to whom study treatment has been assigned by randomization except the additional subjects who were intolerant to the last TKI and were in MMR at baseline.) | 85 | 84 | 0 | 0
Full Analysis Set 2 (FAS 2) (Only the additional subjects who were intolerant to the last TKI and were in MMR at baseline and to whom study treatment has been assigned by randomization.) | 0 | 0 | 14 | 16
Safety Set (SAF) (All subjects who received at least one dose of study treatment except the additional subjects who were intolerant to the last TKI and were in MMR at baseline.) | 84 | 84 | 0 | 0
Safety Set 2 (SAF 2) (Only the additional subjects who were intolerant to the last TKI and achieved were in MMR at baseline and who received at least one dose of study treatment.) | 0 | 0 | 14 | 16
Completed | 0 | 0 | 0 | 0
Not Completed | 85 | 84 | 14 | 16
Not completed — Adverse Event | 6 | 4 | 0 | 2
Not completed — Unsatisfactory Therapeutic Effect | 4 | 3 | 0 | 0
Not completed — Progressive Disease | 1 | 5 | 0 | 0
Not completed — Physician Decision | 2 | 2 | 0 | 0
Not completed — Failure To Meet Continuation Criteria | 2 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Treatment ongoing at the time of the data cut-off date 12-Mar-2024 | 68 | 68 | 14 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Asciminib 40 mg b.i.d. - Subjects Without MMR at Baseline | Asciminib 80 mg q.d. - Subjects Without MMR at Baseline | Asciminib 40 mg b.i.d. - Subjects With MMR at Baseline | Asciminib 80 mg q.d. - Subjects With MMR at Baseline | Total
Number analyzed (Participants) | 85 | 84 | 14 | 16 | 199
Age, Customized [Count of Participants; unit: Participants]
  18 - < 65 years | 64 | 59 | 9 | 11 | 143
  65 - < 75 years | 12 | 19 | 4 | 3 | 38
  >=75 years | 9 | 6 | 1 | 2 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 27 | 6 | 6 | 76
  Male | 48 | 57 | 8 | 10 | 123
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 21 | 21 | 2 | 2 | 46
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 2 | 0 | 0 | 6
  White | 58 | 60 | 12 | 14 | 144
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Major Molecular Response (MMR) Rate at Week 48 for All Patients With no Evidence of MMR at Baseline
Description: Major Molecular Response (MMR) is defined as a significant reduction in the level of BCR::ABL1 transcripts, which are the genetic markers of chronic myeloid leukemia (CML). Specifically, MMR is achieved when there is a ≥ 3.0 log reduction in BCR::ABL1 transcripts compared to a standardized baseline, which corresponds to a BCR::ABL1/ABL1 ratio of ≤ 0.1% on the international scale (IS).
  The Major Molecular Response (MMR) rate at Week 48 for all patients with no evidence of MMR at baseline refers to the percentage of patients who achieve MMR after 48 weeks of treatment, despite not having MMR at the start.
Time Frame: Week 48
Population: Full Analysis Set (FAS)
Measure: Number (95% Confidence Interval); unit: Percentage of responders
Arm/Group | Asciminib 40 mg b.i.d. - Subjects Without MMR at Baseline | Asciminib 80 mg q.d. - Subjects Without MMR at Baseline
Number analyzed (Participants) | 85 | 84
Percentage of responders | 42.35 [31.70 to 53.55] | 34.52 [24.48 to 45.69]

2. Secondary Outcome: MMR Rate at Week 12, 24, 36, 72, 96 and 144 for Patients With no MMR at Baseline
Description: The Major Molecular Response (MMR) rate at alternative time points (weeks 12, 24, 36, 72, 96 and 144) for all patients with no evidence of MMR at baseline refers to the percentage of patients who achieve MMR after those respective weeks of treatment, despite not having MMR at the start. MMR itself is defined as achieving a BCR::ABL1 ratio of ≤ 0.1%.
Time Frame: Week 12, 24, 36, 72, 96 and 144
Reporting Status: Not Posted, anticipated posting 2027-07

3. Secondary Outcome: Major Molecular Response (MMR) Rate at Week 48 for Patients With MMR at Baseline
Description: The Major Molecular Response (MMR) rate at Week 48 for patients with MMR at baseline refers to the percentage of patients who maintain or achieve MMR after 48 weeks of treatment. MMR itself is defined as achieving a BCR::ABL1 ratio of ≤ 0.1%.
Time Frame: Week 48.
Population: Full Analysis Set 2 (FAS 2) and with evaluable data at the pre-specified time points
Measure: Number (95% Confidence Interval); unit: Percentage of responders
Arm/Group | Asciminib 40 mg b.i.d. - Subjects Without MMR at Baseline | Asciminib 80 mg q.d. - Subjects Without MMR at Baseline
Number analyzed (Participants) | 14 | 14
Percentage of responders | 100 [76.84 to 100.00] | 87.5 [61.65 to 98.45]

4. Secondary Outcome: Time to MMR for Subjects Without MMR at Baseline
Description: Time to MMR defined as the time from the date of randomization to the date of the first documented MMR. MMR itself is defined as achieving a BCR::ABL1 ratio of ≤ 0.1%.
Time Frame: From the date of enrollment to the date of first documented MMR, assessed up to 144 weeks
Reporting Status: Not Posted, anticipated posting 2027-07

5. Secondary Outcome: Rate of BCR::ABL1 ≤ 10% for Subjects Without MMR at Baseline
Description: The rate of BCR::ABL1 ≤ 10% refers to the percentage of patients who achieve a BCR::ABL1 level of 10% or lower within the first 48 weeks of treatment.
Time Frame: Week 12, 24, 36 and 48
Population: Full Analysis Set (FAS)
Measure: Number (95% Confidence Interval); unit: Percentage of BCR::ABL1 <= 10%
Arm/Group | Asciminib 40 mg b.i.d. - Subjects Without MMR at Baseline | Asciminib 80 mg q.d. - Subjects Without MMR at Baseline
Number analyzed (Participants) | 85 | 84
Percentage of BCR::ABL1 <= 10%
  Week 12 | 69.4 [58.47 to 78.95] | 81.0 [70.92 to 88.70]
  Week 24 | 72.9 [62.21 to 82.01] | 76.2 [65.65 to 84.81]
  Week 36 | 71.8 [60.96 to 81.00] | 82.1 [72.26 to 89.65]
  Week 48 | 71.8 [60.96 to 81.00] | 78.6 [68.26 to 86.78]

6. Secondary Outcome: Rate of BCR::ABL1 ≤ 1% for Subjects Without MMR at Baseline
Description: The rate of BCR::ABL1 ≤ 1% refers to the percentage of patients who achieve a BCR::ABL1 level of 1% or lower within the first 48 weeks of treatment.
Time Frame: Week 12, 24, 36 and 48.
Population: Full Analysis Set (FAS)
Measure: Number (95% Confidence Interval); unit: Percentage of BCR::ABL1 ≤ 1%
Arm/Group | Asciminib 40 mg b.i.d. - Subjects Without MMR at Baseline | Asciminib 80 mg q.d. - Subjects Without MMR at Baseline
Number analyzed (Participants) | 85 | 84
Percentage of BCR::ABL1 ≤ 1%
  Week 12 | 61.2 [49.99 to 71.56] | 53.6 [42.35 to 64.53]
  Week 24 | 64.7 [53.59 to 74.77] | 58.3 [47.06 to 69.00]
  Week 36 | 63.5 [52.38 to 73.71] | 64.3 [53.08 to 74.45]
  Week 48 | 64.7 [53.59 to 74.77] | 59.5 [48.25 to 70.10]

7. Secondary Outcome: Deep Molecular Responses (MR4) Rate for Subjects Without MMR at Baseline
Description: Deep molecular responses (MR4) is defined as a ≥ 4 log reduction in BCR::ABL1 transcripts compared to the standardized baseline, equivalent to 0.01% BCR::ABL1/ABL1 by the international scale (IS).
Time Frame: Week 12, 24, 36, 48, 72, 96 and 144.
Reporting Status: Not Posted, anticipated posting 2027-07

8. Secondary Outcome: Deep Molecular Responses (MR4.5) Rate for Subjects Without MMR at Baseline
Description: Deep molecular responses (MR4.5) is defined as a ≥ 4.5 log reduction in BCR::ABL1 transcripts compared to the standardized baseline, equivalent to 0.0032% BCR::ABL1/ABL1 by the international scale (IS).
Time Frame: Week 12, 24, 36, 48, 72, 96 and 144.
Reporting Status: Not Posted, anticipated posting 2027-07

9. Secondary Outcome: Rate of Complete Cytogenetic Response (CCyR) for Subjects Without MMR at Baseline
Description: Cytogenetic Response is assessed based on the percentage of Philadelphia chromosome-positive (Ph+) metaphases in the bone marrow, with a review of at least 20 metaphases required.
  Complete Cytogenetic Response (CCyR) is defined as 0% Ph+ metaphases in the bone marrow.
Time Frame: Week 48 and end of treatment (up to 144 weeks)
Reporting Status: Not Posted, anticipated posting 2027-07

10. Secondary Outcome: Occurrence of High-risk Additional Chromosomal Abnormalities (ACA) for Subjects Without MMR at Baseline
Description: High-risk additional chromosomal abnormalities (ACAs) are specific chromosomal abnormalities that are considered to increase the risk in Philadelphia chromosome-positive (Ph+) cells.
Time Frame: Up to 144 weeks
Reporting Status: Not Posted, anticipated posting 2027-07

11. Secondary Outcome: Cumulative Molecular Response Rate of BCR::ABL1 ≤ 10% for Subjects Without MMR at Baseline
Description: The cumulative molecular response rate refers to the proportion of subjects achieving a BCR::ABL1 level of ≤ 10% on the international scale (IS) over a specified period.
Time Frame: From enrollment to end of treatment up to 144 weeks.
Reporting Status: Not Posted, anticipated posting 2027-07

12. Secondary Outcome: Cumulative Molecular Response Rate of BCR::ABL1 ≤1% for Subjects Without MMR at Baseline
Description: The cumulative molecular response rate refers to the proportion of subjects achieving a BCR::ABL1 level of ≤ 1% on the international scale (IS) over a specified period.
Time Frame: From enrollment to end of treatment up to 144 weeks.
Reporting Status: Not Posted, anticipated posting 2027-07

13. Secondary Outcome: Cumulative Molecular Response Rate of MMR for Subjects Without MMR at Baseline
Description: The cumulative molecular response rate refers to the proportion of subjects achieving MMR, defined as a BCR::ABL1 ratio of ≤ 0.1% on the international scale (IS), over a specified period.
Time Frame: From enrollment to end of treatment up to 144 weeks.
Reporting Status: Not Posted, anticipated posting 2027-07

14. Secondary Outcome: Cumulative Molecular Response Rate of MR4 for Subjects Without MMR at Baseline
Description: The cumulative molecular response rate refers to the proportion of subjects achieving MR4, defined as a ≥ 4 log reduction in BCR::ABL1 transcripts compared to the standardized baseline, equivalent to 0.01% BCR::ABL1/ABL1 by the international scale (IS), over a specified period.
Time Frame: From enrollment to end of treatment up to 144 weeks.
Reporting Status: Not Posted, anticipated posting 2027-07

15. Secondary Outcome: Cumulative Molecular Response Rate of MR4.5 for Subjects Without MMR at Baseline
Description: The cumulative molecular response rate refers to the proportion of subjects achieving MR4.5, defined as a ≥ 4.5 log reduction in BCR::ABL1 transcripts compared to the standardized baseline, equivalent to 0.0032% BCR::ABL1/ABL1 by the international scale (IS), over a specified period.
Time Frame: From enrollment to end of treatment up to 144 weeks.
Reporting Status: Not Posted, anticipated posting 2027-07

16. Secondary Outcome: Duration of MMR
Description: Duration of MMR is defined as the time from the date of first documented MMR to the earliest date of loss of MMR, progression to accelerated phase (AP) or blast crisis (BC), or CML-related death. The duration of MMR is analyzed for the subjects in FAS who achieved MMR at any time.
Time Frame: From the date of the first documented molecular response at MMR level to the date of first documented loss of the response level or death due to any cause, whichever occurs first, assessed up to 144 weeks.
Reporting Status: Not Posted, anticipated posting 2027-07

17. Secondary Outcome: Duration of MR4 Without Loss of MMR
Description: Duration of MR4 without loss of MMR refers to the period during which a patient maintains a deep molecular response (MR4) without experiencing a loss of Major Molecular Response (MMR).
Time Frame: From the date of first documented MR4 without loss of MMR to the date of first documented loss of the response level or death due to any cause, whichever occurs first, assessed up to 144 weeks.
Reporting Status: Not Posted, anticipated posting 2027-07

18. Secondary Outcome: Progression-Free Survival (PFS) for Subjects Without MMR at Baseline
Description: Progression-Free Survival (PFS) is defined as the time from the date of randomization to the earliest occurrence of documented disease progression to AP/BC or the date of death from any cause, assessed up to approximately 144 weeks. The time will be censored at the date of last study assessment (PCR, cytogenetic, hematologic or extramedullary) or last post-treatment follow-up for subjects without event. PFS (in months) is calculated as: (date of disease progression/death or censoring date - date of randomization +1)/30.4375.
Time Frame: Up to 144 weeks.
Reporting Status: Not Posted, anticipated posting 2027-07

19. Secondary Outcome: Overall Survival (OS) for Subjects Without MMR at Baseline
Description: Overall Survival (OS) is defined as the time from treatment assignment to death due to any cause during study, assessed up to 144 weeks. Subjects who are alive at the time of the analysis data cutoff date will be censored at the date of last contact before the cut-off date. OS (in months) is calculated as: (date of death or censoring date - date of randomization + 1)/30.4375.
Time Frame: Up to 144 weeks.
Reporting Status: Not Posted, anticipated posting 2027-07

20. Secondary Outcome: Time to Treatment Failure (TTF) for Subjects Without MMR at Baseline
Description: Time from treatment assignment to treatment failure is defined as BCR-ABL1>10%, assessed up to 144 weeks. For subjects who have not reached treatment failure, their TTFs will be censored at the time of last study assessment (PCR, cytogenetic, hematologic or extramedullary) before the cut-off date. TTF (in months) is calculated as: (date of treatment failure or censoring date - date of randomization + 1)/30.4375.
Time Frame: Up to 144 weeks.
Reporting Status: Not Posted, anticipated posting 2027-07

21. Secondary Outcome: Change in Symptom Burden and Interference From Baseline Over Time According to the MDASI-CML PRO Instrument
Description: The MD Anderson Symptom Inventory - Chronic Myeloid Leukemia (MDASI-CML) is a 26 item self-administered questionnaire for adult CML patients. Twenty of the items measure the severity of disease-related symptoms (symptom burden) and are scored from 0 (not present) to 10 (as bad as you can imagine) and 6 items that measure symptom interference with daily life (interference) scored from 0 (did not interfere) to 10 (interfered completely). For symptom burden, total scores range from 0 to 200 and for interference range from 0 to 60, with higher scores indicates high impact on severity of chronic myeloid leukemia-related symptoms and on impact of these symptoms on daily functioning for the patient.
Time Frame: Week 4, 12, 24, 48, 72, 96, 120 and at end of treatment (up to 144 weeks).
Reporting Status: Not Posted, anticipated posting 2027-07

ADVERSE EVENTS:
Time Frame: From first dose of study treatment up to the cut-off date for the Week 48 primary analysis (12-Mar-2024), approximately 29 months.
Description: All-cause Mortality was assessed for all participants enrolled in the study, while Serious and Other Adverse Events were assessed for all participants who received at least one dose of the study medication (Safety Set (SAF) for subjects without MMR at baseline and Safety Set 2 (SAF2) for subjects with MMR at baseline).
Arm/Group | Asciminib 40 mg b.i.d. - Subjects Without MMR at Baseline | Asciminib 80 mg q.d. - Subjects Without MMR at Baseline | Asciminib 40 mg b.i.d. - Subjects With MMR at Baseline | Asciminib 80 mg q.d. - Subjects With MMR at Baseline
All-Cause Mortality (participants affected / at risk) | 0/85 | 1/84 | 0/14 | 0/16
Serious Adverse Events (participants affected / at risk) | 9/84 | 9/84 | 4/14 | 5/16
Other Adverse Events (participants affected / at risk) | 67/84 | 67/84 | 12/14 | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Asciminib 40 mg b.i.d. - Subjects Without MMR at Baseline (N=84) | Asciminib 80 mg q.d. - Subjects Without MMR at Baseline (N=84) | Asciminib 40 mg b.i.d. - Subjects With MMR at Baseline (N=14) | Asciminib 80 mg q.d. - Subjects With MMR at Baseline (N=16)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Hypersplenism (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Blindness unilateral (Eye disorders) | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Dengue fever (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0
Cervicobrachial syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0
Pelvic haematoma (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Asciminib 40 mg b.i.d. - Subjects Without MMR at Baseline (N=84) | Asciminib 80 mg q.d. - Subjects Without MMR at Baseline (N=84) | Asciminib 40 mg b.i.d. - Subjects With MMR at Baseline (N=14) | Asciminib 80 mg q.d. - Subjects With MMR at Baseline (N=16)
Anaemia (Blood and lymphatic system disorders) | 3 | 3 | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 3 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 7 | 7 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 9 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0 | 1
Bundle branch block left (Cardiac disorders) | 1 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Cushingoid (Endocrine disorders) | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 2 | 2 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 5 | 5 | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 4 | 4 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 6 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 7 | 6 | 1 | 4
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2 | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 1 | 2 | 0 | 1
Lip disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 6 | 8 | 0 | 3
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Asthenia (General disorders) | 6 | 2 | 0 | 0
Fatigue (General disorders) | 3 | 12 | 1 | 1
Gait disturbance (General disorders) | 1 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 2 | 3 | 0 | 1
Pain (General disorders) | 1 | 3 | 1 | 0
Pyrexia (General disorders) | 2 | 3 | 0 | 2
Bacteraemia (Infections and infestations) | 0 | 1 | 1 | 0
Bronchitis (Infections and infestations) | 2 | 4 | 0 | 3
COVID-19 (Infections and infestations) | 11 | 9 | 3 | 3
Folliculitis (Infections and infestations) | 1 | 2 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 1
Influenza (Infections and infestations) | 3 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 1 | 0 | 2
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 1
Tracheobronchitis viral (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 5 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 2 | 2 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 9 | 2 | 0 | 1
Amylase increased (Investigations) | 3 | 2 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 8 | 2 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 1 | 0
Blood cholesterol increased (Investigations) | 2 | 1 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 7 | 1 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 1 | 1
Glycosylated haemoglobin increased (Investigations) | 0 | 0 | 0 | 1
High density lipoprotein decreased (Investigations) | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 6 | 7 | 1 | 2
Low density lipoprotein increased (Investigations) | 1 | 0 | 1 | 2
Platelet count decreased (Investigations) | 4 | 6 | 0 | 0
Prothrombin time prolonged (Investigations) | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 3 | 4 | 2 | 0
Weight increased (Investigations) | 2 | 4 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 | 2 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 13 | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 7 | 0 | 2
Gouty tophus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 4 | 2 | 4
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 5 | 1 | 0 | 0
Headache (Nervous system disorders) | 8 | 8 | 2 | 4
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 2 | 2 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 5 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0
Micturition disorder (Renal and urinary disorders) | 0 | 0 | 0 | 1
Penile erythema (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 2 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 7 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Macule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 5 | 3 | 5
Rash (Skin and subcutaneous tissue disorders) | 3 | 5 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 5 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Angiopathy (Vascular disorders) | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 1 | 1
Hot flush (Vascular disorders) | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 6 | 5 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-08-10): https://cdn.clinicaltrials.gov/large-docs/33/NCT04948333/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-16): https://cdn.clinicaltrials.gov/large-docs/33/NCT04948333/SAP_001.pdf